CLINICAL TRIAL: NCT00548457
Title: Endothelial Function in Patients With Ectatic Compared to Normal Coronary Arteries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Pierre Chouraqui, Sheba Medical Center
Other Study IDs: SHEBA-06-4130-PC-CTIL
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Ectasia
Keywords: the function of the endothelium of the arteries in patients suffering from ectatic coronary arteries
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A

SUMMARY:
The aim of this study is to show the frequency of endothelial dysfunction in patients suffering from ectatic coronary arteries as compared to those who have normal coronary arteries. Should this frequency be significant we would recommend initiating conventional treatment in those patients with ectatic coronary arteries as is the practice in patients with endothelial dysfunction without ectatic arteries

ELIGIBILITY:
Inclusion Criteria:

* Ectatic coronary arteries defined by cardiac catheterization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited after passing cardiac catherization and diagnosed as having ectatic arteries.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chouraqui, MD, Study Chair — Sheba Medical Center
Locations (1):
- Heart Institute, Chaim Sheba Medical Center, Tel Litwinsky, Israel